CLINICAL TRIAL: NCT05493098
Title: Effectiveness of Dry Needling for Suboccipital, Levator Scapula, Upper Trapezius, Masseter, Sternocleidomastoid, Splenius Capitis and Cervicis, Temporalis and Frontalis Muscles on Pain and Active Craniocervical Range of Motion in People With Episodic Tension-type Headache
Brief Title: Effectiveness of Dry Needling in People With Episodic Tension-type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1400.30
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Episodic Tension-type Headache
Keywords: dry needling; tension-type headache; myofascial pain syndrome
MeSH Terms: conditions — Tension-Type Headache; Myofascial Pain Syndromes | interventions — Dry Needling; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will include 18 participants with episodic tension-type headache. The treatment will include dry needling of the suboccipital, levator scapula, upper trapezius, masseter, sternocleidomastoid, splenius capitis, and cervicis, frontalis, and temporalis muscles and routine physical therapy. The needles will be inserted to obtain local twitch response, and this process will continue until no more local twitch response occurs in each session. Then the needles will be left in place for 20 minutes. In each session, three muscles from one side will be needled. Routine physical therapy will include information on nature, management, course of episodic tension-type headaches, and Multimodal care that includes craniocervical exercises and postural correction. The treatment will last two weeks, six sessions, three times a week.
  Interventions: Other: dry needling
- Control group (Placebo Comparator): The control group will include 18 participants with episodic tension-type headache. The treatment will include "sham" dry needling of the suboccipital, levator scapula, upper trapezius, masseter, sternocleidomastoid, splenius capitis, and cervicis, frontalis and temporalis muscles and routine physical therapy. The sham dry needling method includes the insertion of the needles subcutaneously and no local twitch response will be obtained. The needles will be left in the place for 20 minutes. In each session, three muscles from one side will be needled. Routine physical therapy will include information on nature, management, course of episodic tension-type headaches, and Multimodal care that includes craniocervical exercises and postural correction. The treatment will last two weeks, six sessions, three times a week.
  Interventions: Other: sham (placebo) dry needling:

INTERVENTIONS:
Other: dry needling — The method of performing the dry needling technique will be based on the methods presented by Dommerholt and Fernandez-de-Las-Penas. One length of sterile, disposable 0.30 mm x 30 mm solid filament needle (Tony, China) will be used. The length of the needle for each participant will be selected based on the size of the participant. The needles will be inserted to obtain local twitch response, and this process will continue until no more Dry needling:
  The method of performing the dry needling technique will be based on the methods presented by Dommerholt and Fernandez-de-Las-Penas. One length of sterile, disposable 0.30 mm x 30 mm solid filament needle (Tony, China) will be used. The length of the needle for each participant will be selected based on the size of the participant. The needles will be inserted to obtain local twitch response, and this process will continue until no more local twitch response occurs in each session. Then the needles will be left in place for 20 minutes.
  Arms: Experimental group
Other: sham (placebo) dry needling: — The sham dry needling method includes the insertion of the needles subcutaneously and no local twitch response will be obtained. The needles will be left in the place for 20 minutes.
  Arms: Control group

SUMMARY:
Tension-type headache is a widespread disorder, with a lifetime prevalence in the general population ranging between 30% and 78%. Tension-type headache also places a financial burden on society and individuals. Myofascial pain can reduce the range of motion and patterns of muscle activation and play an important role in tension-type headache. Based on the previous studies, dry needling can reduce local and referred pain, increase range of motion and improve patterns of muscle activation in patients with myofascial pain syndrome. The effectiveness of dry needling in patients with tension-type headache is not fully known.

Objective: The aim of this study will be to investigate the effectiveness of dry needling on pain, active range of motion, functional disability, and frequency of headache in patients with episodic tension-type headache.

Method: This study will be a double-blind randomized controlled trial. Thirty-six patients with episodic tension-type headache will be randomly divided into two groups: the experimental group (dry needling and routine physical therapy) and the control group (sham dry needling and routine physical therapy). The primary outcomes will be pain intensity and active range of motion of the craniocervical region. Functional disability and frequency of headache will be considered secondary outcomes. Outcomes will be assessed before and one week after the intervention.

DETAILED DESCRIPTION:
Study design: The experimental design will be a randomized, sham-controlled, double-blind, parallel assignment design to investigate the effectiveness of dry needling on pain, active range of motion, functional disability, and frequency of headache in patients with episodic tension-type headache. This investigation will be conducted in the physiotherapy clinic located at the School of Rehabilitation Sciences, Iran University of Medical Sciences, Tehran, Iran. The ethical committee at the Iran University of Medical Sciences has approved this study (Ethical Approval Number: IR.IUMS.REC.1400.30).

Participants: The sample size of this investigation was calculated using Stata statistical software (version 14) with an α value of 0.05 to achieve a statistical power of 0.95 and an effect size of 0.2. The results revealed that a minimum of 36 patients with episodic tension-type headache is required. All of the participants will be identified and recruited by posters and word-of-mouth from the University and the surrounding local communities. Eligible participants will be explained the purpose and the examination involved in this investigation, and all eligible participants will sign a written informed consent before entering the study.

Randomization: All eligible episodic tension-type headache patients will be randomized to an experimental group (dry needling of suboccipital, levator scapula, upper trapezius, masseter, sternocleidomastoid, splenius capitis and cervicis, frontalis and temporalis muscle and routine physical therapy) and a control group (sham dry needling of suboccipital, levator scapula, upper trapezius, masseter, sternocleidomastoid, splenius capitis and cervicis, frontalis and temporalis muscle and routine physical therapy) with a ratio of 1:1. Random allocation will be executed by a researcher not involved in the assessments or interventions. Patients will be asked not to provide their grouping information to the assessor to prevent data contamination.

Procedure: Before the examination, the demographic characteristics form, including name, age, occupation, weight, height, smoking, type and duration of pain, and history of other diseases will be recorded. Primary outcomes are pain level and active range of motion of the craniocervical vertebra.

Functional disability, frequency of headache, and side effects of dry needling are considered secondary outcomes. The numeric pain rating scale, manual goniometer, and neck disability index will be used to measure pain level, active range of motion ,and functional disability, respectively. Outcomes will be examined at baseline and one week after the end of the intervention. Patients will be asked about the side effects of dry needling, such as soreness during and after dry needling, bleeding, etc., at the end of the treatment sessions. The examiner will be blinded to the intervention procedure. Patients will also be blinded to which group they belong to.

Intervention: The intervention will be for six sessions, two weeks, three times a week.

Experimental group: The method of performing the dry needling technique will be based on the methods presented by Dommerholt and Fernandez-de-Las- Penas. In this method, patients will be placed in a supine position for masseter, temporalis, sternocleidomastoid, and frontalis.

Sternocleidomastoid: The Sternocleidomastoid Both heads, clavicular and sternal, will be needled by pincer palpation after identifying the carotid artery. The needle is then inserted perpendicular to the skin and directed towards the practitioner's finger.

Temporalis: The tempolaris muscle will be needled with flat palpation. The needle is fixed with the index and middle fingers of the non-needling hand and then inserted perpendicular to the skin toward the temporalis fossa.

Masseter: The muscle will be needled with flat palpation, although pincer palpation may also be feasible. The needle will be inserted perpendicular to the skin toward the muscle belly.

Frontalis: The frontalis muscle will be needled with flat palpation. The needle will be inserted in oblique and inferior direction, 1 cun above the middle of the eyebrow, directly above the pupil when the eyes are looking straight ahead.

Patients will be placed in the lateral decubitus position for levator scapula, splenius capitis, and cervicis.

Levator scapula: The muscle will be needled via pincer palpation. For the superior (cervical) portion, the muscle is felt as a ropy muscle band of about 5mm diameter in lateral extent, between the anterior (ventral) border of the upper trapezius and the transverse process of C1. The needle will be inserted perpendicular to the skin and directed towards the practitioner's finger. For the lower (shoulder) portion, the muscle is identified over the superior medial border of the scapula. The needle will be inserted through the skin at a shallow angle, directed toward the upper, medial border of the scapula.

Splenius capitis: In splenius capitis, one finger is placed on the taut band. The needle is inserted through the skin at a shallow angle in a caudal-medial direction and directed toward the practitioner's finger.

Splenius cervicis: This muscle will be needled via pincer palpation. The needle will be inserted perpendicular to the skin from a posterior to anterior direction, directed towards the practitioner's finger or at a shallow angle. The needle may be directed medially because the muscle is laterally away from the cervical spine foramina. The needle may be through the upper fibers of the trapezius muscle.

Patients will be placed in a prone position for upper trapezius and suboccipital. Upper trapezius: The muscle will be needled via pincer palpation. The needle will be inserted perpendicular to the skin from a posterior to anterior direction directed towards the practitioner's finger or at a shallow angle. The muscle will be needled with pincer palpation. The needle will be inserted perpendicular to the skin and directed towards the practitioner's finger. The needle is kept between the fingers on the shoulder.

Suboccipital: The muscle will be needled at a point mid-way between the transverse process of C1 and the spinous process of C2. The needle will be inserted perpendicular to the skin directly in the medial half of the muscle toward the patient's opposite eye in a slightly cranial-medial direction.

One length of sterile, disposable 30 mm x 30 mm solid filament needle (Tony, China) will be used. The needles will be inserted to obtain local twitch response,which continues until no more local twitch response occurs in each session. Then the needles will be left in the place for 20 minutes. In each session, the muscles from one side will be needled.

Control group: The sham dry needling method includes inserting the needles subcutaneously and no local twitch response will be obtained. The needles will be left in the place for 20 minutes.

Routine physical therapy will be based on the guideline by Côté et al. (2019) and include information on nature, management, course of episodic tension-type headaches, and Multimodal care that includes craniocervical exercises and postural correction. To give information to patients, we will use the Persian version of tutorials provided by ICHD-3. Multimodel care consists of three exercises: chin tuck, upper trapezius and levator scapula stretch, and pectoralis major stretch. Stretching exercise will be done three times a day, with three repetitions and 30 seconds of hold position. Chin tuck will be done five times a day with ten repetitions.

Outcome measure: Outcomes will be assessed at baseline and one week after the intervention (after six sessions of treatment). The examiner will be blinded to the intervention procedure.

Pain level: The 0-100 Numeric Pain Rating Scale (NPRS) will be used to evaluate changes in the level of pain from the baseline to one week after the intervention. Zero indicates no pain and 100 indicates maximum pain that the patient experiences.

Active Craniocervical range of motion:

Active craniocervical range of motion of participants with episodic tension-type headache will be measured using a SAEHAN plastic universal two-arm goniometer with 360° goniometer face and 30-cm (11.81- in) movable arms. For measuring active flexion, extension, lateral flexion, and rotation, the participants will be asked to sit upright on a chair with a padded backrest supporting the thoracic spine with their feet flat on the floor and arms positioned comfortably on the armrests beside them. To minimize the contribution of the thoracic spine, the participants will be securely strapped across the shoulders to the chair using an inelastic belt. To standardize head posture, a visual target (white A5 paper with a black circle drawn upon it) will be adjusted to eye level in front of the participants. To measure active craniocervical flexion and extension ROM, the center of the universal goniometer will be placed over the external auditory meatus. Then, the proximal arm (fixed arm) will be positioned perpendicular to the floor and the distal arm (moving arm) will be placed over an imaginary line between the base of the nostril and the external auditory meatus. One surface of the universal goniometer face will be covered with a white sheet of paper so that the figures cannot be seen from the examiner's side. Active lateral flexion ROM will be measured by placing the center of the universal goniometer over the spinous process of C7, the proximal arm will be perpendicular to the floor, and the distal arm will be aligned with the occipital protuberance. Finally, to measure active craniocervical left and right rotation ROM, the center of the universal goniometer will be positioned at the center of the head, the proximal arm will be placed over the sagittal suture, and at the end of the movement, the distal arm Will be aligned with the nose. All the measured angles will be documented by a third person. The movements will be measured in the following sequences: flexion, extension, left lateral flexion, right lateral flexion, left rotation, and right rotation.

Functional disability: The Persian version of the neck disability index will be used to evaluate changes in functional disability from the baseline to one week after the intervention. This questionnaire includes ten activities of daily living and a total score of 50.

Frequency of headache: The participants will be given a notebook to write down the number of the days of the month involved in episodic tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CTTH based on the International Classification of Headache Disorders, 3rd edition
2. At least one active trigger point in each of the muscles of the sub occipital, sternocleidomastoid, upper trapezius, temporalis, levator scapula, masseter, frontalis, and splenius cervicis and capitis
3. Moderate pain intensity from 30 to 60 based on the numeric pain rating scale

Exclusion Criteria:

1. Needle phobia
2. History of surgery on head, neck, and shoulder
3. pregnancy
4. cancer, infectious diseases, or systemic diseases
5. History of involvement with other types of primary headaches
6. History of neck radiculopathy and other orthopedic neck injuries (including fractures, facet joint syndrome, etc.) in the past year.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain level | Change between baseline and one week after intervention.
  0-100 Numeric Pain Rating Scale will be used to evaluate changes in level of pain from the baseline to one week after the intervention. Zero indicates no pain and 100 indicates maximum pain that the patient experiences.
Active craniocervical range of motion | Change between baseline and one week after intervention.
  Active craniocervical range of motion of the participants with episodic tension-type headache will be measured using a SAEHAN plastic universal two-arm goniometer with 360° goniometer face and 30-cm (11.81- in) movable arms. For measuring active flexion, extension, lateral flexion, and rotation, the participants will be asked to sit upright on a chair with a padded backrest supporting the thoracic spine with their feet flat on the floor and arms positioned comfortably on the armrests beside them. To minimize the contribution of the thoracic spine, the participant will be securely strapped across the shoulders to the chair using an inelastic belt. All the measured angles will be documented by a third person. The movements will be measured in the following sequences: flexion, extension, left lateral flexion, right lateral flexion, left rotation, and right rotation.

SECONDARY OUTCOMES:
Functional disability | Change between baseline and one week after intervention.
  The Persian version of the neck disability index will be used to evaluate changes in functional disability from the baseline to one week after the intervention. This questionnaire includes 10 activities of daily living and a total score of 50. higher scores indicate a greater degree of disability.
Frequency of headache: | Change between baseline and one week after intervention.
  The participants will be given a notebook to write down the number of days of the month involved in episodic tension-type headaches.

IPD SHARING:
Plan to Share IPD: Yes
The data sets of this study will be available upon a reasonable request to the corresponding author.

REFERENCES:
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Chowdhury D. Tension type headache. Ann Indian Acad Neurol. 2012 Aug;15(Suppl 1):S83-8. doi: 10.4103/0972-2327.100023. PMID 23024570
- [Background] Dowson A. The burden of headache: global and regional prevalence of headache and its impact. Int J Clin Pract Suppl. 2015 May;(182):3-7. doi: 10.1111/ijcp.12650. PMID 25907016
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Fumal A, Schoenen J. Tension-type headache: current research and clinical management. Lancet Neurol. 2008 Jan;7(1):70-83. doi: 10.1016/S1474-4422(07)70325-3. PMID 18093564
- [Background] Bendtsen L. Central sensitization in tension-type headache--possible pathophysiological mechanisms. Cephalalgia. 2000 Jun;20(5):486-508. doi: 10.1046/j.1468-2982.2000.00070.x. PMID 11037746
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Cuadrado ML, Gerwin RD, Pareja JA. Myofascial trigger points and their relationship to headache clinical parameters in chronic tension-type headache. Headache. 2006 Sep;46(8):1264-72. doi: 10.1111/j.1526-4610.2006.00440.x. PMID 16942471
- [Background] Kamonseki DH, Lopes EP, van der Meer HA, Calixtre LB. Effectiveness of manual therapy in patients with tension-type headache. A systematic review and meta-analysis. Disabil Rehabil. 2022 May;44(10):1780-1789. doi: 10.1080/09638288.2020.1813817. Epub 2020 Sep 12. PMID 32924640
- [Background] Cagnie B, Dewitte V, Barbe T, Timmermans F, Delrue N, Meeus M. Physiologic effects of dry needling. Curr Pain Headache Rep. 2013 Aug;17(8):348. doi: 10.1007/s11916-013-0348-5. PMID 23801002
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] Kamali F, Mohamadi M, Fakheri L, Mohammadnejad F. Dry needling versus friction massage to treat tension type headache: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):89-93. doi: 10.1016/j.jbmt.2018.01.009. Epub 2018 Jan 31. PMID 30691768
- [Background] Mousavi SJ, Parnianpour M, Montazeri A, Mehdian H, Karimi A, Abedi M, Ashtiani AA, Mobini B, Hadian MR. Translation and validation study of the Iranian versions of the Neck Disability Index and the Neck Pain and Disability Scale. Spine (Phila Pa 1976). 2007 Dec 15;32(26):E825-31. doi: 10.1097/BRS.0b013e31815ce6dd. PMID 18091478
- [Background] Cote P, Yu H, Shearer HM, Randhawa K, Wong JJ, Mior S, Ameis A, Carroll LJ, Nordin M, Varatharajan S, Sutton D, Southerst D, Jacobs C, Stupar M, Taylor-Vaisey A, Gross DP, Brison RJ, Paulden M, Ammendolia C, Cassidy JD, Loisel P, Marshall S, Bohay RN, Stapleton J, Lacerte M. Non-pharmacological management of persistent headaches associated with neck pain: A clinical practice guideline from the Ontario protocol for traffic injury management (OPTIMa) collaboration. Eur J Pain. 2019 Jul;23(6):1051-1070. doi: 10.1002/ejp.1374. Epub 2019 Feb 28. PMID 30707486
- [Background] Fernandez-de-Las-Penas C, Florencio LL, Plaza-Manzano G, Arias-Buria JL. Clinical Reasoning Behind Non-Pharmacological Interventions for the Management of Headaches: A Narrative Literature Review. Int J Environ Res Public Health. 2020 Jun 9;17(11):4126. doi: 10.3390/ijerph17114126. PMID 32527071
- [Background] van Ettekoven H, Lucas C. Efficacy of physiotherapy including a craniocervical training programme for tension-type headache; a randomized clinical trial. Cephalalgia. 2006 Aug;26(8):983-91. doi: 10.1111/j.1468-2982.2006.01163.x. PMID 16886935
- [Background] Madsen BK, Sogaard K, Andersen LL, Tornoe B, Jensen RH. Efficacy of strength training on tension-type headache: A randomised controlled study. Cephalalgia. 2018 May;38(6):1071-1080. doi: 10.1177/0333102417722521. Epub 2017 Jul 27. PMID 28750588
- [Background] Madsen BK, Sogaard K, Andersen LL, Skotte J, Tornoe B, Jensen RH. Neck/shoulder function in tension-type headache patients and the effect of strength training. J Pain Res. 2018 Feb 23;11:445-454. doi: 10.2147/JPR.S146050. eCollection 2018. PMID 29503581
- [Background] Farooq MN, Mohseni Bandpei MA, Ali M, Khan GA. Reliability of the universal goniometer for assessing active cervical range of motion in asymptomatic healthy persons. Pak J Med Sci. 2016 Mar-Apr;32(2):457-61. doi: 10.12669/pjms.322.8747. PMID 27182261